CLINICAL TRIAL: NCT03342456
Title: The Efficacy and Safety of Ilaprazole/Doxycycline-based Bismuth-containing Quadruple Therapy on Hp Infected Duodenal Ulcers: A Randomized, Parallel-controlled Multi-center Study
Brief Title: The Efficacy and Safety of Ilaprazole/Doxycycline-based Bismuth-containing Quadruple Therapy on Hp Infected Duodenal Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Collaborators: Livzon Pharmaceutical Group Inc. (Industry); Yung Shin Pharm. Ind. Co., Ltd. (Industry)
Responsible Party: Principal Investigator, XU CANXIA, Director, Clinical Professor of Department of Gastroenterology, Principal Investigator, The Third Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: xucanxia2000
Record Dates: First submitted 2017-10-30; First posted 2017-11-17 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Duodenal Ulcer Due to Helicobacter Pylori
Keywords: Helicobacter pylori eradication; Duodenal Ulcer; Ilaprazole/Doxycycline-based Bismuth-containing quadruple therapy
MeSH Terms: conditions — Duodenal Ulcer | interventions — Amoxicillin; Furazolidone; Potassium Citrate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): week1 to week2：Doxycycline Hyclate Enteric-Coated Capsules 0.1g,orally,twice daily,taken with meals, Ilaprazole Enteric-Coated Tablets 5mg,orally,twice daily, Furazolidone Tablets 0.1g,orally,twice daily,taken with meals, Bismuth Potassium Citrate Tablets 220mg,orally,twice daily week3 to week4：Ilaprazole Enteric-Coated Tablets 5mg,orally,once daily
  Interventions: Drug: Doxycycline Hyclate Enteric-Coated Capsules; Drug: Ilaprazole Enteric-Coated Tablets; Drug: Furazolidone Tablets; Drug: Potassium Citrate Tablets
- group 2 (Active Comparator): Amoxicillin Capsules 1g,orally,twice daily,taken with meals, Ilaprazole Enteric-Coated Tablets 5mg,orally,twice daily, Furazolidone Tablets 0.1g,orally,twice daily,taken with meals, Bismuth Potassium Citrate Tablets 220mg,orally,twice daily.
  week3 to week4：Ilaprazole Enteric-Coated Tablets 5mg,orally,once daily
  Interventions: Drug: Amoxicillin Capsules; Drug: Ilaprazole Enteric-Coated Tablets; Drug: Furazolidone Tablets; Drug: Potassium Citrate Tablets

INTERVENTIONS:
Drug: Doxycycline Hyclate Enteric-Coated Capsules — group 1,0.1g*10 capsules/box, produced by Yung Shin Pharm.Ind.(Kunshan) Co.,Ltd.
  Arms: group 1
Drug: Amoxicillin Capsules — group 2,0.5g*24 capsules/box, produced by United Laboratories（Zhuhai）
  Arms: group 2
Drug: Ilaprazole Enteric-Coated Tablets — group 1 and group 2,5mg*6 capsules/box, produced by Livzon Pharmaceutical Group Inc
Drug: Furazolidone Tablets — group 1 and group 2,0.1g*100 tablets/bottle,produced by Shanxi Yunpeng Pharmaceutical co.,Ltd.
Drug: Potassium Citrate Tablets — group 1 and group 2,110mg*40 tablets/bottle,produced by Livzon Pharmaceutical Group Inc

SUMMARY:
Helicobacter pylori (Hp) infection is one of the important causes of gastrointestinal diseases, including gastritis, peptic ulcer, and malignancies, nd the eradication of Hp can effectively cure or prevent these diseases. Now, owing to the increasingly serious antibiotic resistance, Hp eradication rate is, however, becoming decreased. In order to improve the eradication rate of Hp, clinicians pay great attention to choose more effective treatment.

Ilaprazole Enteric-Coated Tablets is a new generation of proton pump inhibitor (PPI). Previous research found that Ilaprazole had a more prolonged half-life and higher suppression of gastric acid secretion. In addition, its metabolism is not significantly influenced by CYP2C19, compared to the available PPIs. Doxycycline is in the tetracycline antibiotic class, has a stronger antibacterial force than tetracycline and its antibacterial spectrum is basically the same as tetracycline and doxycycline, so far, it is not widely used. Preliminary observations showed that Ilaprazole/Doxycycline-based quadruple therapy was effective in treating Hp infection, with less adverse reactions and good compliance with patients.

In this study, a multi-center, randomized, parallel controlled trial will be conducted in 7 hospitals in Hunan Province, China, to observe the clinical efficacy and safety of the Bismuth-containing quadruple therapy with Ilaprazole, Doxycycline, Furazolidone and Bismuth Potassium Citrate in the treatment of Hp infected duodenal ulcer. It is expected to complete 200 effective cases, including 100 cases in the experimental group and 100 cases in the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Has endoscopic evidence of active duodenal ulcer(within a week before participate), accompanying or not accompanied with abdominal pain/abdominal discomfort, acid, heartburn, abdominal distention, belching and other corresponding symptoms.
2. The diameter of the ulcer is 0.3 to 2.0cm, and the number is less than or equal 2.
3. Has evidence(s) of Hp infection. (13C-UBT/14C-UBT/Pathological test)
4. Has a history of antiacid medication, but has been stopped for more than 2 weeks.
5. Has not used antibiotics and (or) bismuth agents in nearly four weeks.
6. Understand and be willing to participate in this clinical trial.

Exclusion Criteria:

1. Has been taking ulcer medications, such as non-steroidal anti-inflammatory drugs, adrenal corticosteroids etc.
2. Has allergic and idiosyncratic responses to the tested drugs and (or) control drugs.
3. Has a diagnosis of duodenal carcinelcosis or a duodenal ulcer can not rule out the the possibility of malignancy (patients with gastrointestinal mucosal epithelial mild atypical hyperplasia are not ruled out) or compound ulcers.
4. Has severe or progressive dysphagia, weight loss, gastrointestinal bleeding or other alarm symptoms.
5. Has esophageal or gastric varices, Zollinger-Ellison syndrome, or serious complications such as pyloric obstruction, active bleeding in the endoscope; esophageal erosion or ulcers, other digestive serious diseases, Such as Crohn's disease, ulcerative colitis.
6. Has a history of gastric acid suppression surgery, esophageal surgery, or digestive organ surgery, with the exception of simple suture of perforation.
7. Is pregnant, breastfeeding or has a family planning during whole trail.
8. Has serious cardiovascular, pulmonary, hepatic, renal, hematological or endocrine disease with uncontrolled condition.
9. Has participated in other clinical trials within 3 months prior to the trial.
10. Is required to use the prescribed anti-ulcer drug during the trial.
11. Has a history of drug and (or) alcohol abuse.
12. Has restriction on sodium, with metabolic alkalosis and (or) hypocalcemia.
13. Has a long-term use of clopidogrel.
14. Has other reasons for not to participating in clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
The eradication rate of H. pylori infection | Visit period 3 (After day 56)
  Evaluated by 13C-urea breath test (13C-UBT), 14C-urea breath test (14C-UBT), or Pathological examination.

SECONDARY OUTCOMES:
The healing rate of duodenal ulcer(s) | Visit period 2 (day 28±1)
  Duodenal ulcer healing rate is defined as the percentage of participants with complete healing of ulcer (according to Sakita-Fukutomi classification) under endoscope.
Number of duodenal ulcer(s) | Visit period 2 (day 28±1)
  Confirmed by endoscope.
Maximum diameter of duodenal ulcer(s) | Visit period 2 (day 28±1)
  Confirmed by endoscope (cm).
Surrounding inflammation and(or) erosion of duodenal ulcer(s) | Visit period 2 (day 28±1)
  Confirmed by endoscope.
Incidence of bleeding | Visit period 2 (day 28±1)
  Confirmed by endoscope.
Improvement of gastric symptoms | Screening period (day -3~0), Visit period 1 (day 14±1), Visit period 2 (day 28±1)
  Improvement is defined as the total change from baseline symptoms scores of Symptom Rating Scale(Includidng 9 items: Pain in day, Pain in night, Burning in day, Burning in night, Acid reflux in day, Acid reflux in night, Nausea and vomiting, Belching, Abdominal distension. Depending on severity and frequency, scale ranges from 0-3 points.).

OTHER OUTCOMES:
Degree of pain | Screening period (day -3~0), Visit period 1 (day 14±1), Visit period 2 (day 28±1)
  Evaluated by clinical symptoms scores
  1. Pain in day 0 point: No pain. 1 point: Mild pain, do not affect daily life and work, do not have to take medicines. 2 points: Obvious pain,partly affect daily life and work, or have to take medicines. 3 points: Severe pain, must rest, taking medicine is ineffective
  2. Pain in night 0 point: No pain. 1 point: Mild pain, do not affect daily life and work, do not have to take medicines. 2 points: Obvious pain,partly affect daily life and work, or have to take medicines. 3 points: Severe pain, must rest, taking medicine or eat is ineffective
Degree of burning | Screening period (day -3~0), Visit period 1 (day 14±1), Visit period 2 (day 28±1)
  Evaluated by clinical symptoms scores
  1. Burning in day 0 point: No burning. 1 point: Occasionally. 2 points: Frequently and duration prolonged. 3 points: Continuously, use antacid to alleviate briefly.
  2. Burning in night 0 point: No burning. 1 point: Occasionally. 2 points: Frequently and duration prolonged. 3 points: Continuously, use antacid to alleviate briefly.
Degree of acid reflux | Screening period (day -3~0), Visit period 1 (day 14±1), Visit period 2 (day 28±1)
  Evaluated by clinical symptoms scores
  1. Acid reflux in day 0 point: No acid reflux. 1 point: Occasionally. 2 points: One to two times a day. 3 points: Several times a day.
  2. Acid reflux in night 0 point: No acid reflux. 1 point: Occasionally. 2 points: One to two times a day. 3 points: Several times a day.
Degree of nausea and vomiting | Screening period (day -3~0), Visit period 1 (day 14±1), Visit period 2 (day 28±1)
  Evaluated by clinical symptoms scores Nausea and vomiting 0 point: No nausea. 1 point: Occasionally and briefly. 2 points: Frequent nausea, vomiting. 3 points: Continuous nausea, frequent vomiting.
Degree of belching | Screening period (day -3~0), Visit period 1 (day 14±1), Visit period 2 (day 28±1)
  Evaluated by clinical symptoms scores Belching 0 point: No belching. 1 point: Occasionally. 2 points: Frequently. 3 points: Continuously, and affect normal activities.
Degree of abdominal distension | Screening period (day -3~0), Visit period 1 (day 14±1), Visit period 2 (day 28±1)
  Evaluated by clinical symptoms scores Abdominal distension 0 point: No abdominal distension. 1 point: Occasionally. 2 points: Obvious abdominal distension. 3 points: Severe abdominal distension, and affect normal activities.
Symptom disappearance time | Visit period 1 (day 14±1), Visit period 2 (day 28±1)

CONTACTS AND LOCATIONS:
Overall Officials: JINGSHU CHI, Principal Investigator — The Third Xiangya Hospital of Central South University; XIAOMING LIU, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (7):
- China (7):
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - Loudi central hospital, Loudi, Hunan
  - Shaoyang Central Hospital, Shaoyang, Hunan
  - The Affiliated Hospital Of YongZhou Vocational Technical College, Yongzhou, Hunan

IPD SHARING:
Plan to Share IPD: No